CLINICAL TRIAL: NCT00964626
Title: A Phase II Study of Efficacy and Safety of Paclitaxel and Cisplatin Every 2 Weeks as the First-line Treatment of Patients With Ovarian Cancer Stage Ic-IV.
Brief Title: Paclitaxel and Cisplatin as First-Line Treatment for Patients With Stage I, Stage II, Stage III, or Stage IV Ovarian Epithelial Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Russian Academy of Medical Sciences (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000641288; USSR-AMS-PAC-2; EU-20937; BIOCAD-PAC-2
Record Dates: First submitted 2009-08-22; First posted 2009-08-25 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Ovarian Cancer
Keywords: stage IA ovarian epithelial cancer; stage IB ovarian epithelial cancer; stage IC ovarian epithelial cancer; stage IIA ovarian epithelial cancer; stage IIB ovarian epithelial cancer; stage IIC ovarian epithelial cancer; stage IIIA ovarian epithelial cancer; stage IIIB ovarian epithelial cancer; stage IIIC ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Cisplatin; Paclitaxel

INTERVENTIONS:
Drug: cisplatin
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects of giving paclitaxel together with cisplatin as first-line therapy and to see how well it works in treating patients with stage I, stage II, stage III, or stage IV ovarian epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To investigate the efficacy and safety of paclitaxel and cisplatin as first-line chemotherapy in patients with stage IC-IV ovarian epithelial cancer.

OUTLINE: This is a multicenter study.

Patients receive paclitaxel IV and cisplatin IV once every 2 weeks. Treatment repeats every 2 weeks for 9 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed epithelial adenocarcinoma of the ovary

  * Stage IC-IV disease
* No known or clinical evidence of brain metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Hemoglobin must be ≥ 90 g/L
* ANC ≥ 2 x 10^9/L
* Platelet count ≥ 100 x10^9/L
* Serum creatinine ≤ 115 μmol/L
* Total bilirubin ≤ 25 μmol/L
* Not pregnant or nursing
* No other serious disease which could affect protocol compliance and results
* No other prior malignancy within the past 5 years except for curatively treated carcinoma in situ of the cervix or squamous carcinoma of the skin
* No peripheral neuropathy ≥ CTCAE version 3.0 grade 2
* No known hypersensitivity to any of the study drugs or their excipients
* No drug addiction or alcoholism
* No disorder which leads to the condition that contraindicates the use of the investigational drugs, or that may affect the patient's compliance with the study requirements

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy for ovarian cancer

Ages: 18 Years to 72 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Overall survival
Objective response rate (complete and partial remission in patients with measurable disease)
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Sergei A. Tjulandin, MD, PhD, Principal Investigator — Russian Academy of Medical Sciences
Locations (1):
- Russian Academy of Medical Sciences Cancer Research Center, Moscow, Russia